CLINICAL TRIAL: NCT05891210
Title: Nutritional Assessment in Children With Congenital Heart Disease
Brief Title: Nutrition in Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanaa Atia Mohamed Hasanin, Nutritional assessment in children with congenital heart disease, Assiut University
Other Study IDs: congenital heart
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease (CHD) defined as anatomic malformation of the heart and great vessels which occurs during intrauterine development irrespective of the age of presentation(1) It is classified into acyanotic and cyanotic depending upon whether the patients clinically exhibit cyanosis(2) .

It is the most common human developmental anomaly with a reported prevalence of between 4 to 10 per 1000 live birth (3-6).

The variety and severity of clinical presentation depend on the cardiac structures involved and their functional impact (7).

Previous studies have found that, although birth weight for gestational age is usually normal in patients with congenital heart disease, young children often present with impaired growth parameters (8,9) The underlying causes of this failure to thrive may be multifactorial including innate growth potential, severity of cardiac underlying disease, increased energy requirements ,decreased nutritional intake, malabsorption and poor utilization of absorbed nutrients .these factor are particularly common and sever in low and middle income countries (11) Several studies suggest that the failure to thrive is associated with poorer cognitive development, learning disabilities, and long term behavioral problems more recently Corbett et al (12) detected a significant association between the severity of growth deficiency and IQ ,whereas Raynor and Rudolf (13) found that 55% of the infants who were failing to thrive exhibited developmental delay .In addition , A study by Reif et al (14) reported that children with a history of failure to thrive were found to have more learning difficulties and evidenced developmental delay at follow up 5 years after the initial presentation(15).

Achieving survival is not the only target of clinicians for these patients, appropriate growth, development and improved quality of life are also very important.

The management of children with congenital heart disease require multidisciplinary approach,in which the nutritional aspect plays an important role ,an adequate caloric intake, in fact this improve the out come of these patients.(7) This study will asses the nutritional status for patients with congenital heart disease Who are admitted at assiut university hospital children and adopting a protocol for nutritional support for them.

DETAILED DESCRIPTION:
1. Full history taking including date of birth,gender,residence,and socioeconomic status.

   According To Socioeconomic status we will ask about where the family live,family income (high or middle or low income) Perinatal history as maternal age,gestational diseases,medications use during pregnancy,irradiation exposure ,presence of antenatal care.

   Natal hisrory ;mode of delivery(vainal,cesarean) ,site of delivery (home,hospital) Post natal history; required resuscitation or not,cyanosis,jaundice and incubator care needed or not,birth weight will be categorized into appropriate ,small or large for gestational age.

   Feeding history; breast or formula feeding,age of weaning ,type of food for weaning, supplementation of vitamin D.iron.
2. All patients will subject to general and systemic examination. Children included in our study will fall under Complete general and systemic examination especially heart disease.
3. Nutritional assessment and anthropometric measures will be followed up to these patients; AThe weight ; will be taken on a scale that has been properly calibrated and the value will be plotted on a standardized WHO growth chart .

B)The height ; this measurement for children more than 2years will be taken without shoes using astadiometer and the value will be plotted on the WHO growth chart.

C)The length; this measurement in children 2 years and younger is more accurate ,the child will position in supine on ameasuring board.

D)Head circumference; will be measured using a flexible tabe ,we will measure the maximum diameter through the supraorbital ridge to the occiput and the value will be plotted on the growth chart.

E)Mid arm circumference; this measured using a flexible nonstretch tape laid at the midpoint between the acromion and olecranonprocesses on the shoulder blade and the ulna respectively.

F) BMI:

Measured by the person's weight divided by the square of height in meters for children aged more than 2years and will be plotted at the WHO growth chart.

ELIGIBILITY:
Inclusion Criteria:

* Children more than one month and till age of 18 years that present to Assiut University Hospital Units with Cyanotic and ACyanotic Congenital heart disease will be included in our study.

Exclusion Criteria:

* All pediatric patients with comorbidities other than congenital heart disease will be excluded from our study as: severe sepsis, endocarditis, empyema& autoimmune diseases& liver cirrhosis& children receiving immunosuppressive therapy

Ages: 5 Weeks to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children more than one month and till age of 18 years that present to Assiut University Hospital Units with Cyanotic and ACyanotic Congenital heart disease will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Asses the nutritional status of the children with congenital heart disease | Baseline
  Adopt a protocol to avoid nutritional deficiency and achieve the normal growth in children with congenital heart disease.